CLINICAL TRIAL: NCT02586467
Title: Testing the Effectiveness of Targeted, Framed, -Efficacy Enhancing Messages for Increasing Milk and Milk Product Consumption in Adults Aged 30--50 Years.
Brief Title: Messages for Increasing Dairy Consumption
Acronym: MilkMessage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mary Jung, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H12-00332
Record Dates: First submitted 2015-10-20; First posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Gain-Framed (Experimental): Participants receive messages that highlight the potential benefits of engaging in a specific behaviour (i.e., what positive outcomes they could experience from consuming milk and milk products).
  Interventions: Behavioral: Gain-Framed
- Loss-Framed (Experimental): Participants receive messages that highlight the potentially loses of not engaging in a specific behaviour (i.e., what they could lose from not consuming milk and milk products).
  Interventions: Behavioral: Loss-Framed
- Self-Regulatory Efficacy (Experimental): Participants receive messages that provide them with tips and strategies on how to engage in the consumption of milk and milk products (i.e., recipes, meal planning etc.)
  Interventions: Behavioral: Self-Regulatory Efficacy
- Gain-Framed + Self-Regulatory Efficacy (Experimental): Participants receive messages that highlight the potential benefits of engaging in a specific behaviour (i.e., what positive outcomes they could experience from consuming milk and milk products) and these messages also provide tips and strategies on how to engage in the consumption of milk and milk products (i.e., recipes, meal planning etc.).
  Interventions: Behavioral: Gain-Framed + Self-Regulatory Efficacy
- Loss-Framed + Self-Regulatory Efficacy (Experimental): Participants receive messages that highlight the potentially loses of not engaging in a specific behaviour (i.e., what they could lose from not consuming milk and milk products) and these messages also provide tips and strategies on how to engage in the consumption of milk and milk products (i.e., recipes, meal planning etc.).
  Interventions: Behavioral: Loss-Framed + Self-Regulatory Efficacy

INTERVENTIONS:
Behavioral: Gain-Framed — Participants will be randomised to one of five message conditions. Each condition will receive a total of four emailed messages on four consecutive days (i.e., 1 message per day). Participants in the Gain-Framed message condition will receive message content that highlights the potential benefits of consuming milk and milk products (i.e., high protein content, stronger hair and nail etc.)
  Arms: Gain-Framed
Behavioral: Loss-Framed — Participants will be randomised to one of five message conditions. Each condition will receive a total of four emailed messages on four consecutive days (i.e., 1 message per day). Participants in the Loss-Framed message condition will receive message content that highlights the potential losses of not consuming milk and milk products (i.e., lack of essential nutrients, less calcium).
  Arms: Loss-Framed
Behavioral: Self-Regulatory Efficacy — Participants will be randomised to one of five message conditions. Each condition will receive a total of four emailed messages on four consecutive days (i.e., 1 message per day). Participants in the Self-Regulatory Efficacy message condition will receive information pertaining to how to include milk and milk products within their diet. This information will come in the form of recipes, meal planning, food combining etc.
  Arms: Self-Regulatory Efficacy
Behavioral: Gain-Framed + Self-Regulatory Efficacy — Participants will be randomised to one of five message conditions. Each condition will receive a total of four emailed messages on four consecutive days (i.e., 1 message per day). Participants in the Gain-Framed message + Self-Regulatory Efficacy condition will receive message content that highlights the potential benefits of consuming milk and milk products (i.e., high protein content, stronger hair and nail etc.) and information pertaining to how to include milk and milk products within their diet.
  Arms: Gain-Framed + Self-Regulatory Efficacy
Behavioral: Loss-Framed + Self-Regulatory Efficacy — Participants will be randomised to one of five message conditions. Each condition will receive a total of four emailed messages on four consecutive days (i.e., 1 message per day). Participants in the Loss-Framed message + Self-Regulatory Efficacy condition will receive message content that highlights the potential losses of not consuming milk and milk products (i.e., lack of essential nutrients, less calcium) and information pertaining to how to include milk and milk products within their diet.
  Arms: Loss-Framed + Self-Regulatory Efficacy

SUMMARY:
Over 35,000 Canadians, 65% of men and 72% of women aged 31-50 years fail to consume the recommended number of milk and milk product servings (≤2 servings per day). Given the wide range of health benefits associated with increased dietary intake of milk and milk products the objectives of this study were to conduct a prospective, 5-arm randomised controlled trial in order to test the effectiveness of a variety of messages for increasing milk and milk product consumption in men and women aged 30-50 years old. The five arms consisted of 4 messages that contained slightly different content specifically: 1) gain-framed message condition, 2) loss-framed message condition, 3) self-regulatory efficacy-enhancing message condition, 4) gain-framed and self-regulatory efficacy-enhancing message condition and 5) loss-framed plus self-regulatory efficacy-enhancing message condition. It was hypothesised that those who receive self-regulatory efficacy-enhancing information would consume more dairy than those who received messages without such information. Second, those who received gain-framed messages would consume more dairy as compared to those who received loss-framed messages. Third, those who received gain-framed messages that include self-regulatory efficacy-enhancing information would consume the most dairy in comparison to the other four conditions.

ELIGIBILITY:
Inclusion Criteria:

* Between 30 and 50 years of age
* Consume less than 2 servings of milk or milk products per day
* No health or religious reasons to avoid milk and milk products
* Regular access to the internet
* Can speak and read English

Exclusion Criteria:

* Dietary restrictions, allergies, or medical reasons for limiting dairy intake will be excluded

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 732 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in calcium from dairy at 1 and 4-week follow up | Baseline, 1-week follow-up, 4-week follow-up
  Calcium consumed from dairy was assessed using a modified version of the "Calcium Calculator™" developed by the British Columbia Dairy Foundation. The original tool assesses consumption of calcium from a comprehensive list of 30 commonly consumed calcium containing products. For this study individuals were asked to indicate the portions they ate of 10 dairy products included in the list. An explanation of a portion was provided for each item. Milligrams of calcium consumed by participants on the previous day was determined for baseline, week 1 and week 4 follow-up.

SECONDARY OUTCOMES:
Self-Regulatory Efficacy | Baseline, Immedately after the Intervention (1-day), 4-Week Follow-Up
  Changes in participants self-regulatory efficacy beliefs was assessed using an 18-item measure at baseline, 1-day after completion of the intervention and at 4-week follow-up. Self-regulatory efficacy beliefs items were context specific. Responses were scored on a scale of 0% (not at all) to 100% (extremely confident) with response options in 10% increments.
Outcome Expectations | Baseline, Immedately after the Intervention (1-day), 4-Week Follow-Up
  Changes in participants outcome expectations was assessed at baseline, 1-day after completion of the intervention and at 4-week follow-up. The perceived likelihood of positive (16 items) and negative (5 items) outcomes occurring as a result of consuming milk and milk products was assessed using a 21-item measure. Responses were scored on a 9-point scale from 1 (very unlikely) to 9 (very likely).
Outcome Values | Baseline, Immedately after the Intervention (1-day), 4-Week Follow-Up
  Changes in participants outcome values was assessed at baseline, 1-day after completion of the intervention and at 4-week follow-up. The perceived value of positive (16 items) and negative (5 items) outcomes occurring as a result of consuming milk and milk products was assessed using a 21-item measure. Responses were scored on a 9-point scale with a range of 1 (little value to me) to 9 (high value to me).

CONTACTS AND LOCATIONS:
Locations (1):
- Health and Exercise Psychology Laboratory, Kelowna, British Columbia, Canada

REFERENCES:
- [Background] Tversky A, Kahneman D. The framing of decisions and the psychology of choice. Science. 1981 Jan 30;211(4481):453-8. doi: 10.1126/science.7455683.
- [Background] Jung ME, Martin Ginis KA, Phillips SM, Lordon CD. Increasing calcium intake in young women through gain-framed, targeted messages: a randomised controlled trial. Psychol Health. 2011 May;26(5):531-47. doi: 10.1080/08870441003611544. PMID 21557134
- [Background] Bandura A. Social foundations of thought and action: A social cognitive theory. NJ US: Prentice-Hall, Inc; 1986.